CLINICAL TRIAL: NCT06082154
Title: A Prognostic Model Based on POCUS at ICU Admission in Critically Ill Patients With Sepsis
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Ashmita Paudel, Principal Investigator, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 506(6-11)E2
Record Dates: First submitted 2023-10-07; First posted 2023-10-13 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-08

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — Patient will undergo multiorgan ultrasonography

SUMMARY:
Sepsis is responsible for one in three patient deaths. Understanding the severity of the disease, directing medications, prognosticating, and communicating with family members depend on the ability to predict outcomes in a patient presenting with sepsis in the ICU. The outcome of mortality reflects the caliber of ICU treatment. This is a prospective observational study that will include all patients diagnosed with sepsis for point-of-care ultrasonography within 24 hours of admission to the ICU from April 26, 2023, to March 30, 2024, and create a model that will predict 28 day outcome in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Age >=16 yrs within 24 hour of ICU admission diagnosed as Sepsis as per Sepsis 3

Exclusion Criteria:

* USG cannot be done within 24 hour of admission to icu If USG cannot be done for 2 parameters Who do not give consent Withdrawal of active life support Do not intubate(DNI) or do not resuscitate(DNR) order at admission

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient who are diagnosed as having sepsis as per Sepsis 3 definition
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
28 day status alive or dead | 28 days
  patient will be followed for 28 days from day of icu admission to find out their status being alive or dead

CONTACTS AND LOCATIONS:
Locations (1):
- Ashmita Paudel, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No